CLINICAL TRIAL: NCT00698750
Title: A Prospective, Non-controlled, Clinical Investigation of the Copeland™ Humeral Resurfacing Head
Brief Title: A Clinical Investigation of the Copeland™ Humeral Resurfacing Head
Status: Terminated | Type: Observational
Why Stopped: Sponsor terminated study early due to limited enrollment and follow-up.
Sponsor: Biomet Orthopedics, LLC (Industry)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Other Study IDs: Biomet 12381-30
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Avascular Necrosis; Humeral Fractures
Keywords: Fractured Humeral Head; Traumatic Arthritis; Resurfacing Shoulder; Shoulder Replacement; Shoulder Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Osteonecrosis; Humeral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Copeland™ Humeral Resurfacing Head: Copeland™ Humeral Resurfacing Head

SUMMARY:
The purpose of this study is to perform a five-year, prospective evaluation of the Copeland™ Humeral Resurfacing Head Prosthesis for outcome and durability. Relief of pain and restoration of function will determine long-term clinical outcome while durability will be measured by the absence of revisions.

ELIGIBILITY:
Inclusion Criteria:

* Non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis.
* Rheumatoid arthritis
* Correction of functional deformity
* Reconstructable Rotator Cuff
* Treatment of acute fracture of the humeral head
* Traumatic arthritis

Exclusion Criteria:

* Patients less than 18 years.
* Patients with rapid joint destruction, osteomalacia, osteoporosis, or marked bone loss, which would preclude proper fixation of the prosthesis.
* Patients with marked bone loss apparent on roentgenogram.
* Metabolic disorders, which may impair bone formation.
* Patients who are pregnant.
* Patients with an active or suspected infection in or around the shoulder or distant foci of infections, which may spread to the implant site.
* Patients with severe instability or deformity of the ligaments and/or surrounding soft tissue, which would prelude stability of the prosthesis.
* Patients who have had revision procedures where other devices or treatments have failed.
* Patients with a highly communicable disease or diseases that may limit follow-up (e.g. immuno-compromised conditions, hepatitis, active tuberculosis, neoplastic disease, etc).
* Patients unwilling or unable to comply with a rehabilitation program for a cemented or cementless partial or total shoulder replacement or who indicate difficulty or inability to return for follow-up visits prescribed by the study protocol.
* Patients with previous shoulder surgery or conditions that may interfere with the partial or total shoulder replacement's survival or outcome.
* Patients who qualify for inclusion in the study, but refuse consent to participate in the study.
* Patients who have had a partial or total shoulder arthroplasty on the contralateral shoulder within the last year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring humeral resurfacing.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2004-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
ASES Assessment | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years
X-rays | 6 months, 1 year, 2 years, 3 years, 4 years, 5 years

SECONDARY OUTCOMES:
Incidence of revision or removals | Any time

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Beres, MD, Study Director — Director, Clinical Research, Biomet Orthopedics, LLC